CLINICAL TRIAL: NCT00631722
Title: Multicenter, Open-Label, Randomised, Haloperidol-controlled Study to Evaluate Seroquel as Mono-Therapy in the Treatment of Agitated Symptoms in the Patients With Acute Episode of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Si Tianmei, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443C00011
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2008-02

CONDITIONS: Schizophrenia
Keywords: PANSS; Acute Episode of Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Quatiapine Fumarate
- B (Active Comparator)
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Quatiapine Fumarate — 600-750mg/day
  Arms: A
Drug: Haloperidol — 12-20mg/day
  Arms: B

SUMMARY:
This study attempts to observe the efficacy (response time) and safety of the second-generation antipsychotic agent-quetiapine versus the first-generation antipsychotic agent-haloperidol, in treating acute schizophrenia episode and to evaluate the effect of the effectiveness of acute schizophrenia episode on long-term tolerability.

DETAILED DESCRIPTION:
Both medication and patient can affect the compliance of patients to treatment. The control of schizophrenia syndromes effectively and rapidly will build up the confidence of patients on treatments. These early effects may influence the long-term compliance and prognosis of patients. And the antipsychotic medications with neuroprotection effect can significantly improve the long-term prognosis of patients, too.In the past, we always think that there is "delayed onset of antipsychotic" by antipsychotic medications. Recently, a large sample study indicated that the onset of antipsychotic effect was as early as the first day after administration (in 24 hours). This study was carried out in order to compare the second-generation antipsychotic agent- quetiapine with the first-generation antipsychotic agent- haloperidol on the onset time of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided by legal guardians and/or patients.
2. Age from 18-60 years old (inclusion), male or female, inpatients or outpatients.
3. A diagnosis of schizophrenia by ICD-10 criteria as F20.0, F20.1, F20.2 and F20.3.
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment.
5. Able to understand and comply with the requirements of the study.
6. PANSS total score at least 60 with EC factor score at least 15 at both screening and randomisation.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Diagnosis of other mental disorders including mood disorder, schizoform disorder, schizoaffective disorder, delusional disorder, transient psychotic disorder etc.
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others.
4. Known intolerance or lack of response to quetiapine fumarate and haloperidol, as judged by the investigator.
5. Known lack of response to clozapine, as judged by the investigator.
6. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir.
7. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids.
8. Within one dosing interval for long acting antipsychoticsUse.
9. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by ICD-10 criteria.
10. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by ICD-10 criteria within 28 days prior to enrolment.
11. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment.
12. Unstable or inadequately treated medical illness (e.g. CHF - congestive heart failure, angina pectoris, hypertension) as judged by the investigator.
13. Involvement in the planning and conduct of the study.
14. Previous enrolment or randomisation of treatment in the present study.
15. Participation in another drug trial within 28 days prior enrolment into this study or longer in accordance with local requirements.
16. Use of antipsychotics 2 days prior to study treatment
17. Use of clozapine 28 days prior to study treatment.
18. Use of ECT 1 months prior to screening.
19. Initiate quetiapine or haloperidol treatment within 30 days prior to screening.
20. Use of MAOI 14 days prior to study treatment
21. The patient's complete blood count (CBC) with white blood cell (WBC) differential shows an neurotrophil count of ≤ 1.5 x 109/L at screening
22. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) >8.5%
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks
    * Not under physician care for DM
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled
    * Physician responsible for patient's DM care has not approved patient's participation in the study
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to allocation to treatment. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the onset of action quetiapine fumarate (seroquel) in the treatment of Chinese schizophrenic patient with agitation compared with haloperidol by the analysis of time to reduction of PANSS-EC by 20 % | 28 days

SECONDARY OUTCOMES:
To evaluate the global efficacy of seroquel in the treatment of schizophrenia patient with agitation compared with haloperidol by evaluation of change of PANSS total score and CGI-S score from baseline to Week 4 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Tianmei Si, MD, Principal Investigator — Mental Health Institute of Peking University